CLINICAL TRIAL: NCT00151333
Title: A Randomized, Double-blind, Placebo-controlled, Safety, Tolerability, Pharmacokinetics, Pharmacodynamics Trial of Multiple Ascending Fixed Doses of SRA-333 in Subjects With Mild to Moderate Alzheimer's Disease.
Brief Title: Study Evaluating SRA-333 in Mild to Moderate Alzheimer's Disease (AD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3098A1-200
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

INTERVENTIONS:
Drug: SRA-333

SUMMARY:
To determine the safety and tolerability of multiple ascending fixed oral doses of SRA-333 in subjects with mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD according to the NINCDS-ADRDA criteria.
* Men and postmenopausal or surgically sterile women aged from 50 to 85 inclusive.
* Able to give informed consent. Patient's caregiver must consent to participate in the study.

Exclusion Criteria:

* Significant neurologic disease other than AD that may affect cognition.
* Current clinically significant systemic illness which is likely to deteriorate or affect the subject's safety during the study.

Other exclusions apply

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16
Dates: Start 2005-02; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of multiple ascending fixed oral dose in subject with mild to moderate Alzheimer's Disease

SECONDARY OUTCOMES:
To assess the pharmacokinetics and pharmacodynamics of multiple ascending fixed dose.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (3):
- United States (3):
  - Phoenix, Arizona
  - Fort Lauderdale, Florida
  - Miami, Florida